CLINICAL TRIAL: NCT05404256
Title: Randomized Controlled Trial for Comparison of the Effects of Preventing Postoperative Pancreatic Fistula by With Versus Without TissuePatchTM Cover the Wound Surface of Pancreatic Capsule
Brief Title: Comparison of Effectiveness of TissuePatchTM in Preventing Postoperative Pancreatic Fistula
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Xijing Hospital of Digestive Diseases (Other)
Responsible Party: Principal Investigator, xiaohua li, Associate chief physician, Xijing Hospital of Digestive Diseases
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: XJ013
Record Dates: First submitted 2022-05-30; First posted 2022-06-03 (Actual); Last update posted 2024-05-08 (Actual); Status verified 2024-05

CONDITIONS: Pancreatic Fistula
Keywords: TissuePatchTM; radical gastrectomy; postoperative pancreatic fistula
MeSH Terms: conditions — Pancreatic Fistula

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- The experimental group (Experimental): Radical gastrectomy +D2 lymphadenectomy +TissuePatchTM to seal pancreatic tissue surface
  Interventions: Other: Radical gastrectomy +D2 lymphadenectomy+TissuePatchTM to seal pancreatic tissue surface
- The control group (Other): Radical gastrectomy +D2 lymphadenectomy
  Interventions: Other: Radical gastrectomy +D2 lymphadenectomy

INTERVENTIONS:
Other: Radical gastrectomy +D2 lymphadenectomy+TissuePatchTM to seal pancreatic tissue surface — Radical gastrectomy +D2 lymphadenectomy+TissuePatchTM to seal pancreatic tissue surface
  Arms: The experimental group
Other: Radical gastrectomy +D2 lymphadenectomy — Radical gastrectomy +D2 lymphadenectomy
  Arms: The control group

SUMMARY:
Postoperative pancreatic fistula is one of the most serious complications after gastric cancer surgery and can lead to surgery-related death. Postoperative pancreatic fistula for gastric cancer often occurs in accidental injury of pancreas during peripancreatic lymph node dissection, blunt separation of pancreatic capsule injury, laparoscopic instrument clamp and long-term compression of pancreas, etc. TissePatchTM is a synthetic, self-adhesive, absorbable surgical sealant and barrier used to seal and reinforce wounds and prevent leakage of air, blood, and fluid during neurosurgery, spine, chest, and soft tissue surgery. Therefore, we proposed whether the use of TissuePatchTM can reduce the occurrence of pancreatic fistula after gastric cancer surgery, and the clinical trial of the effectiveness of TissuePatchTM on the prevention of pancreatic fistula after radical gastrectomy of gastric cancer can provide new clinical data for the prevention of pancreatic fistula after gastric cancer surgery, and help reduce a series of adverse reactions caused by pancreatic fistula in patients.

DETAILED DESCRIPTION:
Gastric cancer is the fifth most common tumor and the fourth most deadly cancer disease in the world. Surgical resection is the recommended method to cure gastric cancer. In recent years, with the continuous promotion of D2 radical gastrectomy and the rapid development of new technologies such as laparoscopic and robotic surgical systems, although the incidence of complications such as abdominal bleeding, anastomotic leakage and abdominal infection has decreased, but the incidence of Postoperative pancreatic fistula is increasing. Postoperative pancreatic fistula involves the delivery of any measurable volume of fluid through surgically placed drainage tubes, and amylase activity is 3 times higher than the upper limit of normal plasma value. According to the severity of postoperative pancreatic fistula, there are three grades: A, B and C. Grade A pancreatic fistula is mainly biochemical leak (BL), not pancreatic fistula in the real sense. Grade B pancreatic fistula requires a definite change in postoperative treatment strategy, which affects the postoperative process. Continuous drainage of drainage tube in situ for > 3 weeks, or percutaneous or subultrasonic drainage is required; Grade C pancreatic fistula refers to the situation of secondary surgery, single or multiple organ failure (especially respiratory, cardiac and renal insufficiency) and even death caused by postoperative pancreatic fistula. The risk factors of pancreatic fistula after radical gastrectomy for gastric cancer mainly include: 1. Surgical methods and instrument-related factors, such as the scope of surgical resection and lymph node dissection; 2. Pancreatic factors, soft pancreas showed less fibrous tissue, inflammatory cells infiltrating pancreatic tissue and pancreatic edema, and pancreatic fistula was more likely to occur during surgery; 3. Basic information of the patient: obesity is an important risk factor for pancreatic fistula. Currently, laparoscopic surgery has been widely carried out in gastric cancer, but due to the characteristics of laparoscopic surgery and the difference in operator experience, the incidence of postoperative pancreatic fistula is higher than that of open surgery. Postoperative pancreatic fistula is one of the most serious complications after gastric cancer surgery and can lead to surgery-related death. Postoperative pancreatic fistula for gastric cancer often occurs in accidental injury of pancreas during peripancreatic lymph node dissection, blunt separation of pancreatic capsule injury, laparoscopic instrument clamp and long-term compression of pancreas, etc. Due to the digestion of pancreatic fluid, severe pancreatic fistula is often followed by abdominal infection, postoperative bleeding, anastomotic fistula and other serious complications, even life-threatening. Therefore, the prevention and early detection of pancreatic fistula after radical gastrectomy of gastric cancer is very important. At present, there are few studies on the prevention of pancreatic fistula after gastric cancer surgery at home and abroad. The main preventive surgeries require surgeons to perform fine operations and also require individual drainage methods. These methods can reduce the occurrence of pancreatic fistula after gastric cancer surgery to a certain extent, but have weak preventive effect on the large scope of lymph node dissection. TissuePatchTM is a synthetic, self-adhesive, absorbable surgical sealant and barrier used to seal and reinforce wounds and prevent air, blood, and fluid leakage during neurosurgery, spine, chest, and soft tissue surgery. It is a pre-formed patch with built-in adhesive strength. It also incorporates TissuebondTM, a bio-bonding polymer that forms strong covalent bonds to protein-rich tissue surfaces. Adhesion is achieved when the prefabricated membrane is applied to the tissue bed with moderate pressure of 60 seconds, which allows contact adhesion and eliminates potential tissue space. Studies have shown that the use of TissuePatchTM in major neck surgery can effectively prevent the occurrence of chylous leakage and promote the recovery of patients. Therefore, we proposed whether the use of TissuePatchTM can reduce the occurrence of pancreatic fistula after gastric cancer surgery, and the clinical trial of the effectiveness of TissuePatchTM on the prevention of pancreatic fistula after radical gastrectomy of gastric cancer can provide new clinical data for the prevention of pancreatic fistula after gastric cancer surgery, and help reduce a series of adverse reactions caused by pancreatic fistula in patients. Therefore, based on our experience and foundation in the treatment of gastric cancer in gastrointestinal surgery, the real world observation and research on the experimental treatment plan for the prevention of pancreatic fistula in gastric cancer patients after surgery will be carried out, and the integration of domestic superior resources will surely further promote the development of the prevention of pancreatic fistula after radical gastrectomy for gastric cancer.

ELIGIBILITY:
Inclusion Criteria:

* Histological confirmation of gastric adenocarcinoma
* Stage cT1-4a, N0-3, M0 (according to the 8th AJCC TNM staging system)
* For locally advanced tumors (cT3-4aN+M0), preoperative completion of all three cycles of chemotherapy (SOX)
* 18-75 years old
* No incurable factors such as cancer cell metastasis in other organs
* Written informed consent signed voluntarily

Exclusion Criteria:

* Assessment of preoperative or intraoperative requiring pancreatic resection
* Gastric cancer-related emergency surgery
* Gastric stump carcinoma
* In cases of distant metastasis discovered during operation, only abdominal exploration or palliative surgery were adopt.
* Uncontrolled seizures, central nervous system diseases or mental disorders
* Uncorrectable coagulation dysfunction
* Severe uncontrolled recurrent infections or other severe uncontrolled concomitant diseases
* Diseases requiring immunosuppressive treatment, such as organ transplantation, SLE, etc
* Other diseases requiring simultaneous surgery

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 154 (Estimated)
Dates: Start 2022-08-01 (Actual); Primary Completion 2025-04-01 (Estimated); Study Completion 2026-04-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of pancreatic fistula after radical gastrectomy | 3 days
  Postoperative pancreatic fistula, in which any measurable volume of fluid is delivered through a surgically placed drainage tube, has amylase activity greater than 3 times the upper limit of normal plasma value

SECONDARY OUTCOMES:
the postoperative mortality | 30 days
  Postoperative mortality refers to the probability of death within 30 days after radical surgery for gastric cancer
length of postoperative hospital stay | Up to 30 days
  Postoperative hospital stay refers to the time between the date of operation and the date of discharge
Classification of pancreatic fistula | 3 days
  The classification of pancreatic fistula included the incidence of biochemical fistula, grade B pancreatic fistula and grade C pancreatic fistula.
number of lymph nodes dissection | 1 days
  The number of lymph nodes dissected refers to the total number of lymph nodes dissected during the operation
incidence of postoperative complications | 30 days
  incidence of postoperative complications
incidence of TissuePatchTM related complications | 30 days
  intestinal adhesion, intestinal obstruction, parenchymal atrophy of the pancreas, chronic pancreatitis, and allergic reactions and so on.

CONTACTS AND LOCATIONS:
Overall Officials: xiaohua li, MD,PH.D, Study Chair — Xijing Hospital
Locations (1):
- Xijing Hospital of Digestive Disease, Xi'an, Shaanxi, China

REFERENCES:
- [Derived] Yue C, Mo Z, Yang Q, Yu P, Zhou H, Gao R, Wang W, Guo Z, Zhang C, Wang Y, Ji P, Wu X, Zhang Y, Ji G, Li X. Comparison of the efficacy of TissuePatch versus no TissuePatch to seal pancreatic tissue surface for the prevention of pancreatic fistula after radical gastrectomy: study protocol for a prospective, single-center, randomized controlled trial. Trials. 2025 Dec 28. doi: 10.1186/s13063-025-09144-7. Online ahead of print. PMID 41456003